CLINICAL TRIAL: NCT07273110
Title: Effectiveness of Extracorporeal Shock Wave Therapy in Patellofemoral Pain Syndrome: A Randomized Controlled Trial
Brief Title: Extracorporeal Shock Wave Therapy in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uğur Can Yalaki (Other)
Responsible Party: Sponsor-Investigator, Uğur Can Yalaki, MD, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFPS-ESWT-2021
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; extracorporeal shock-wave therapy; exercise therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Active Comparator): Participants performed a structured home-based exercise program targeting hip and knee musculature. The program included warm-up, stretching, and progressive strengthening exercises for the quadriceps, hip abductors, hip external rotators, and core stability muscles. Participants were instructed to complete the program at least three times per week for 4 weeks. Exercise technique and progression guidelines were explained in person, and adherence was monitored using weekly exercise diaries and telephone follow-up.
  Interventions: Behavioral: Home-based Exercise Program
- ESWT (Experimental): Participants received five sessions of radial extracorporeal shock wave therapy (ESWT) administered at 5-day intervals. Treatment was delivered using the Chattanooga Intelect® RPW device with 2000 pulses per session at 1.8-2.0 bar pressure and 8 Hz frequency. Stimulation was applied to the peripatellar soft tissues, including the medial and lateral patellofemoral retinaculum and the infrapatellar fat pad, while avoiding direct application over the patellar tendon. Pressure was progressively increased across sessions based on tolerance.
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy (ESWT)
- Exercise + ESWT (Experimental): Participants performed the same home-based strengthening program as the Exercise group (hip and knee strengthening, ≥3 sessions/week for 4 weeks). In addition, they received five sessions of radial extracorporeal shock wave therapy (2000 pulses; 1.8-2.0 bar; 8 Hz) at 5-day intervals applied to the peripatellar soft tissues while avoiding the patellar tendon.
  Interventions: Behavioral: Home-based Exercise Program; Device: Radial Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Behavioral: Home-based Exercise Program — A structured home-based exercise program targeting hip and knee musculature. The program included warm-up, stretching, and progressive strengthening for the quadriceps, hip abductors, hip external rotators, and core stability muscles. Participants were instructed to perform the program at least three times per week for 4 weeks. Exercise progression and technique were explained individually. Adherence was monitored with weekly exercise diaries and telephone follow-up.
  Arms: Exercise; Exercise + ESWT
Device: Radial Extracorporeal Shock Wave Therapy (ESWT) — Five sessions of radial extracorporeal shock wave therapy delivered at 5-day intervals using the Chattanooga Intelect® RPW device. Each session consisted of 2000 pulses at 1.8-2.0 bar pressure and 8 Hz frequency. Treatment was applied to the peripatellar soft tissues (medial and lateral retinaculum and infrapatellar fat pad), while avoiding direct application over the patellar tendon. Pressure was adjusted based on participant tolerance.
  Arms: ESWT; Exercise + ESWT

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common cause of anterior knee pain and functional limitations in physically active individuals. Exercise-based rehabilitation is considered the primary treatment approach, yet a proportion of patients experience persistent symptoms. Extracorporeal shock wave therapy (ESWT) is a non-invasive modality that may reduce pain through neuromodulation and tissue-level biological responses.

This randomized controlled trial evaluated the effects of ESWT on knee pain and function in adults with PFPS. Thirty-six participants aged 18-45 years were randomly assigned to one of three groups: Exercise, Exercise plus ESWT, or ESWT alone. The exercise program consisted of home-based hip and knee strengthening performed at least three times per week for four weeks. ESWT was administered as five radial shock wave sessions at five-day intervals around the peripatellar soft tissues.

Outcomes included worst knee pain measured by the Visual Analogue Scale and functional status measured by the Kujala Patellofemoral Score at baseline, week 1, and week 8. All groups demonstrated significant improvements over time, with no significant differences between groups. The treatment was well tolerated.

This trial was retrospectively registered after patient enrollment was completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years.
* Clinical diagnosis of patellofemoral pain syndrome (PFPS) characterized by anterior or retropatellar knee pain lasting at least 8 weeks.
* Pain provoked during at least two of the following activities: running, jumping, squatting, stair climbing, or prolonged sitting.
* Worst knee pain score of ≥3 on the Visual Analog Scale (0-10).
* Ability to understand and follow the exercise program and assessment procedures.
* Provided written informed consent.

Exclusion Criteria:

* Evidence of intra-articular knee pathology other than grade 1-2 meniscal changes or grade 1 chondromalacia patella on MRI.
* Clinical signs of patellar instability.
* Localized tenderness indicating alternative diagnoses (e.g., patellar tendinopathy, iliotibial band syndrome, pes anserine bursitis).
* History of knee surgery on the affected side.
* Intra-articular injections (e.g., corticosteroids, hyaluronic acid, PRP) within the past 6 months.
* Neurological or rheumatological disorders affecting the lower extremity.
* Active infection, open wound, tumor, or severe dermatological condition at or near the ESWT application site.
* Pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale, 0-10 | Baseline, Week 1, Week 8
  The Visual Analog Scale (VAS) was used to assess the worst knee pain experienced in the previous week during daily or functional activities. Participants rated their pain on a 0-10 scale, where 0 represents no pain and 10 represents the worst imaginable pain. Pain intensity was recorded at baseline prior to intervention, at one week, and at eight weeks after the treatment to evaluate short- and mid-term treatment effects.

SECONDARY OUTCOMES:
Kujala Patellofemoral Score | Baseline, Week 1, Week 8
  The Kujala Anterior Knee Pain Scale was used to evaluate knee-specific functional status. This validated questionnaire consists of 13 items assessing pain, functional limitations, and activities such as running, stair climbing, prolonged sitting, and squatting. Total scores range from 0 to 100, with higher scores indicating better function. Assessments were completed at baseline, at one week, and at eight weeks after the treatment to determine functional improvement over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ University Sports Medicine Clinic, Bursa, Nilüfer, Turkey (Türkiye)